CLINICAL TRIAL: NCT02287220
Title: Non Contact Measurement of Vital Signs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Robert Thiele, MD, Assistant Professor, Anesthesiology, University of Virginia
Other Study IDs: 17492
Record Dates: First submitted 2014-11-05; First posted 2014-11-10 (Estimated); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Hypoxemia; Hypoxia
Keywords: Non-Contact Oximetry; video plethysmography; oxygen desaturation
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Newborn Infants: 0-12 months old Male or female Any ethnicity
  Interventions: Device: Non-Contact Oximetry

INTERVENTIONS:
Device: Non-Contact Oximetry — Video Record subject when subjected to small amounts of near infrared light

SUMMARY:
The purpose of this study is to test the accuracy of a web cam-based biomedical device developed at UVA (not FDA-approved) that is designed to measure heart rate, respiratory rate, and oxygen saturation without requiring any patient contact. One potential application of such a device would be in the field of infant monitoring allowing parents (and physicians) to monitor the vital signs of infants continuously. The investigators therefore propose to record the heart rate, respiratory rate, and oxygen saturation of 100 infants (defined as children aged 12 months or less) who are receiving continuous oxygen, heart rate, and respiratory rate monitoring with a traditional vital signs monitor. The relationship between "non-contact" and "gold standard" (GE monitoring equipment) heart rate, respiratory rate, and oxygen saturation will be analyzed using regression and limits of agreement analysis.

DETAILED DESCRIPTION:
While multiple investigators have attempted to develop non-contact pulse oximeters, none of these devices have achieved accuracy sufficient for clinical use, no such devices have been approved by the Food and Drug Administration, and there are currently no such devices on the market in the United States. While these devices are typically able to measure the heart and respiratory rates with some accuracy,v the accurate calculation of oxygen saturation from the arterial pulse (SpO2) using a "non-contact" reflectance oximetry probe is complicated by the interference of ambient light, patient temperature changes, as well as the inherent limitations of the sensing devices currently utilized. Poh et al have been somewhat successful at calculating the heart rate from a video recording using independent component analysis. However, Poh's method does not calculate instantaneous rates and requires a facial recognition component to track the facial orientation in the image, is not capable of measuring respiratory rate, and relies primarily on analysis of reflected green light (which cannot be used for the calculation of oxygen saturation). Our work involves modifying a commercial off the shelf (COTS) 3-channel (red, green, blue) CCD (charge coupled device) or CMOS (complementary metal oxide semiconductor) camera in the form of a web cam to detect near infrared and infrared spectrum radiation and applying an algorithm based fast Fourier transformation (FFT) of individual red pixel intensity to detect motion and color changes. Because our algorithm analyzes the first derivative of red pixel intensity, a face-tracking component is unnecessary, and we are able to calculate the heart rate and the respiratory rate in real time.

ELIGIBILITY:
Inclusion Criteria:

* Infant aged 0 - 12 months
* Receiving care at UVA
* Heart rate, respiratory rate, and oxygenation (SpO2) being monitored continuously

Exclusion Criteria:

* Greater than 12 months of age
* Not receiving continuous monitoring of heart rate, respiratory rate, and oxygenation (SpO2) Intubated and/or mechanically ventilated History of retinopathy of prematurity Inability to directly visualize the child's head
* Family unwilling to consent Parents less than 18 years of age

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborn infants that are prone to desaturation events
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2014-11; Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Measure oxygen saturation to be correlated with oxygen saturation calculated from the video recording | 6 hours maximum
  the pulse oximeter saturation will be used as the reference oximeter reading that will be used to validate the oxygen saturation calculated from the video recording
Measure heart rate to be correlated with heart rate calculated from the video recording | 6 hours maximum
  the pulse oximeter heart rate measurement will be used as the reference oximeter reading that will be used to validate the heart rate calculated from the video recording
Measure respiratory rate to be correlated with respiratory rate calculated from the video recording | 6 hours maximum
  the respiratory rate as recorded in the ventilator will be used to validate the respiratory rate calculated from the video recording

CONTACTS AND LOCATIONS:
Overall Officials: Robert Thiele, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sun Y, Papin C, Azorin-Peris V, Kalawsky R, Greenwald S, Hu S. Use of ambient light in remote photoplethysmographic systems: comparison between a high-performance camera and a low-cost webcam. J Biomed Opt. 2012 Mar;17(3):037005. doi: 10.1117/1.JBO.17.3.037005. PMID 22502577
- [Background] Wieringa FP, Mastik F, van der Steen AF. Contactless multiple wavelength photoplethysmographic imaging: a first step toward "SpO2 camera" technology. Ann Biomed Eng. 2005 Aug;33(8):1034-41. doi: 10.1007/s10439-005-5763-2. PMID 16133912
- [Background] Poh MZ, McDuff DJ, Picard RW. Non-contact, automated cardiac pulse measurements using video imaging and blind source separation. Opt Express. 2010 May 10;18(10):10762-74. doi: 10.1364/OE.18.010762. PMID 20588929
- [Background] Verkruysse W, Svaasand LO, Nelson JS. Remote plethysmographic imaging using ambient light. Opt Express. 2008 Dec 22;16(26):21434-45. doi: 10.1364/oe.16.021434. PMID 19104573